CLINICAL TRIAL: NCT06600620
Title: Intelligent Monitoring to Predict Atrial Fibrillation [NOTE-AF]: Clinical Study 1 for the "Health Virtual Twins for the Personalised Management of Stroke Related to Atrial Fibrillation (TARGET)" Project
Brief Title: Intelligent Monitoring to Predict Atrial Fibrillation
Acronym: NOTE-AF
Status: Suspended | Type: Observational
Why Stopped: logistical issues
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: University of Copenhagen (Other); Isansys Lifecare LTD (Unknown); University of Liverpool (Other); Liverpool John Moores University (Other)
Responsible Party: Sponsor
Other Study IDs: JRO-0126
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation New Onset; Postoperative Cardiovascular Complications; Atrial Fibrillation
Keywords: atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (7):
- Patients admitted or referred to Critical Care (NOTE-AF ICU): Patients admitted or referred to Critical Care
  Interventions: Device: Monitoring patients heart rythms with a wireless patch device
- Patients admitted to hospital with acute heart failure (NOTE-AF HF): Patients admitted to hospital with acute heart failure
  Interventions: Device: Monitoring patients heart rythms with a wireless patch device
- Patients admitted to Emergency Services with sepsis or infection (NOTE-AF Sepsis): Patients admitted to Emergency Services with sepsis or infection
  Interventions: Device: Monitoring patients heart rythms with a wireless patch device
- Patients post upper gastrointestinal surgery (NOTE-AF PULSE-GI): Patients post upper gastrointestinal surgery
  Interventions: Device: Monitoring patients heart rythms with a wireless patch device
- Patients post vascular interventions (NOTE-AF Vasc): Patients post vascular interventions
  Interventions: Device: Monitoring patients heart rythms with a wireless patch device
- Patients with acute respiratory failure (NOTE-AF Resp): Patients with acute respiratory failure
  Interventions: Device: Monitoring patients heart rythms with a wireless patch device
- Patients admitted after acute stroke (NOTE-AF stroke): Patients admitted after acute stroke
  Interventions: Device: Monitoring patients heart rythms with a wireless patch device

INTERVENTIONS:
Device: Monitoring patients heart rythms with a wireless patch device — The investigators will collect data in patients at high risk of atrial fibrillation (AF) without a known history of AF to determine clinical predicators of AF. This data will be used to generate virtual digital twins to to predict clinical and subclinical episodes of AF

SUMMARY:
Atrial Fibrillation (AF) is the commonest arrhythmia worldwide, affects 5% of people over the age of 65 and increases the risk of stroke and heart failure. The investigators aim to detect clinical and subclinical episodes of atrial fibrillation lasting >30 seconds to develop risk prediction models to identify patients at high risk for ischaemic stroke.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is the commonest arrhythmia worldwide, affects 5% of people over the age of 65 and increases the risk of stroke and heart failure. Among acutely unwell patients; arrhythmias and myocardial injury are common and associated with increased mortality, morbidity, and healthcare costs. Cardiovascular comorbidities in these high-risk patients include hypertension (47%), dyslipidaemia (29%) and ischaemic heart disease (11%).

The investigators aim to detect clinical and subclinical episodes of atrial fibrillation lasting 30 seconds to develop risk prediction models to identify patients at high risk for ischaemic stroke. Data will serve to develop and validate bedside clinical decision support tools and digital twins. Patients who develop episodes of AF as part of acute illness, will suffer further episodes of AF within one year in over 20% of cases with 27% progressing to paroxysmal/permanent AF. The true incidence of AF is unknown in acutely unwell patients as a significant percentage of AF episodes remain undetected with conventional intermittent monitoring. Patients experiencing short self-terminating episodes of AF carry a 5-fold risk of developing continuous AF and double the risk of stroke and thromboembolic events. Patients suffering episodes of AF often remain asymptomatic but are at increased risk of heart failure and death at one year. Compared to routine intermittent manual measurement of vital signs, wireless continuous vital sign monitoring systems (wCVSM) detect deviations instantaneously with the option of alerting clinical staff in real time via mobile phone applications. Accurate categorization of alerts into false and true events is essential for developing intelligent software that can be embedded into monitoring systems. Continuous ECG and vital signs monitoring can detect AF episodes more reliable, trigger timely investigations and support longer term treatment plans.

Changes in patient pathways and introduction of novel devices to alert healthcare staff on the potential of clinical events require buy-in from all stakeholders. It is therefore essential to evaluate user acceptance and to determine perceptions of users before rolling out a novel patient pathways or implementation of a new device within an organization. The investigators therefore wish to explore users' views of the device, wearing the device and potential areas for improvement using questionnaires for patients and health care staff and by conducting semi-structured interviews with healthcare staff.

Primary objective To determine the true cardiovascular event rate (defined as at least one of the following criteria: episodes of AF, New Regional Wall Motion Abnormalities, raised cardiac biomarkers hs-troponin T and NT-pro-BNP) versus false cardiovascular events detected by continuous wireless remote monitoring.

Secondary objective To determine patient acceptability and usability for health care professionals of a novel remote monitoring device with automated alert function.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥50 years
* Estimated risk of developing new episodes of AF greater than 5%
* Sinus rhythm at presentation
* One of the following acute conditions:

  * Patients admitted or referred to Critical Care (NOTE-AF ICU)
  * Patients admitted to hospital with acute heart failure (NOTE-AF HF)
  * Patients admitted to Emergency Services with sepsis or infection (NOTE-AF Sepsis)
  * Patients post upper gastrointestinal surgery (NOTE-AF PULSE-GI)
  * Patients post vascular interventions (NOTE-AF Vasc)
  * Patients with acute respiratory failure (NOTE-AF Resp)
  * Patients admitted after acute stroke (NOTE-AF stroke)

Exclusion Criteria:

* Atrial fibrillation or atrial flutter at the time of screening
* Patients in atrial fibrillation or atrial flutter at time of preoperative assessment or admission to hospital
* Paced cardiac rhythm
* Inability to obtain consent
* Allergy to plaster or silicone
* Expected hospital stay less than 48 hours

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to hospital with a variety of medical conditions
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence of clinical and subclinical episodes of AF in acutely unwell patients and to generate data for the development and validation of virtual twins and clinical decision support tools. | 48 months
  1) Number of participants with device detected AF lasting greater than 30 seconds
To determine the incidence of clinical and subclinical episodes of AF in acutely unwell patients and to generate data for the development and validation of virtual twins and clinical decision support tools. | 48 months
  Number of episodes of AF and duration of each AF episode

SECONDARY OUTCOMES:
Length of hospital stay | 48 months
  As measured in days and hours
Hospital readmissions within 90 days | 48 months
  Number of readmissions and admission diagnosis of hospital readmissions
Recurrence of AF episodes | 48 months
  Recurrence of AF post discharge as gathered from primary care and secondary care records.
Hospital and 90-day Mortality | 48 months
  Inhospital and 90-day mortality
Time spent in AF | 48 months
  Length of time in AF whilst on monitoring device
Number of AF episodes | 48 months
  Number of AF episodes whilst on monitoring device
Complications of AF | 48 months
  Inhospital and 90 day complications of AF such as stroke, thromboembolic disease & heart failure
High sensitivity Troponin concentrations in patients with AF episodes | 48 months
  Troponin changes (measured by Hs-Trop T) in patients with episodes of AF
Echocardiographic changes in patients with AF episodes | 48 months
  As measured by advanced echocardiographic parameters including but not limited to left atrial conduit strain, left atrial booster strain, left atrial stiffness and left atrial strain
mHealth App Usability Questionnaire | 48 months
  MAUQ score of patients with wireless observations
Percentage change of troponin concentrations in patients with and without episodes of AF | 48 months
  Change in troponin levels in patients with and without episodes of AF
Time wireless continuous vital signs monitoring device is attached | 48 months
  Measured in hours and minutes
Number of cardiovascular alerts | 48 months
  Number of cardiovascular alerts registered by device
Number of non-cardiovascular alerts | 48 months
  Number of non-cardiovascular alerts registered by device
Number of alerts reflecting clinical changes | 48 months
  Number of alerts via continuous vital signs monitoring device
Number of alerts reflecting artefacts or non-clinical events | 48 months
  Number of alerts reflecting clinical deterriorations versus number of alerts reflecting clinical deterrioation
RWMA score, atrial size and volume, left ventricular strain rate, standard echocardiographic measurements as per british society of echocardiography recommendations | 48 months
  Echocardiographic predictors of AF
Change in inflammatory markers white cell count, C-reactive protein and procalcitonin over time | 48 months
  Change in blood tests in patients with and without new-onset AF

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Liverpool university foundation trust, Liverpool
  - Liverpool University hospital Foundation trust, Liverpool

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this point in time

REFERENCES:
- [Derived] Essa H, Johnston B, Lip GYH, Ortega-Martorell S, Williams K, Welters ID; TARGET Consortium. Intelligent monitoring to predict atrial fibrillation (NOTE-AF): clinical study 1 for the 'Health virtual twins for the personalised management of stroke related to atrial fibrillation (TARGET)' project - a protocol for a prospective cohort analysis. BMJ Open. 2026 Jan 3;16(1):e099658. doi: 10.1136/bmjopen-2025-099658. PMID 41485778